CLINICAL TRIAL: NCT00223353
Title: Quantitative Gait Analysis for Clinical Decision Making
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: 978-0011-149
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Joint Disease; Musculoskeletal Equilibrium
Keywords: Biomechanics; Gait; Balance
MeSH Terms: conditions — Joint Diseases | interventions — Braces; Physical Therapy Modalities

GROUPS / COHORTS (2):
- Lower Limb Amputee
  Interventions: Other: Prosthetics, Orthotics and Physical Therapy
- Amputee and Normals and Clinical Case Study: Amputee:
  Lower limb below/above knee amputee
  Normals:
  Health adult
  Clinical Case Study:
  Individual case studies
  Interventions: Other: Prosthetics, Orthotics and Physical Therapy

INTERVENTIONS:
Other: Prosthetics, Orthotics and Physical Therapy — Gait Analysis.

SUMMARY:
The overall purpose of this study is to develop an improved gait analysis system for the real time acquisition, calculation and interpretation of joint kinematic and kinetic information using linked segment body model animation to display and visually depict deviations from normal motion and joint function.

Patients referred to the laboratory for clinical gait analysis are invited to participate in the project. If interested, subjects are informed by a study investigator of the study goals, procedures, risks and any benefits. A study investigator is responsible for obtaining informed consent. Data from normal subjects are used to establish a normative database. Data from other subjects contributes to the relevant databases of different disorders.

DETAILED DESCRIPTION:
The overall purpose of this study is to develop an improved gait analysis system for the real time acquisition, calculation and interpretation of joint kinematic and kinetic information using linked segment body model animation to display and visually depict deviations from normal motion and joint function.

Subjects will be studied using the standard protocol used for patient evaluations in the Rehabilitation Medicine Human Motion Laboratory (GBO13 V AH). The standard protocol includes the routine collection of kinematic data, kinetic data, foot pressure data and, in selected cases, electromyography information. All collected raw data will ultimately be processed for relevant biomechanical parameters and utilized to build either a Normative Database or Non-Normative Database from which selected cases maybe extracted for teaching purposes, pilot data or software development. The project is not designed to test specific hypothesis and as such statistical analysis are not planned.

To acquire kinematics data, infrared reflective markers are taped over the joints of the lower extremities, trunk, and arms. The reflective markers are used in conjunction with the optoelectronic kinematic motion analysis system (Vicon) to allow acquisition of 3D motion data for the limb and trunk segments of subjects. Joint kinetics are determine from ground reaction forces measured by force plates embedded into the floor of the gait laboratory and requiring no specific subject setup. Foot pressure data is obtained by Fscan. Mylar pressure sensitive strips are placed in the shoe or residual limb. The strip is connected to a datalogger and battery pack that will be put on a belt and worn over the shoulder or on the waist. When electromyographic data is required, surface electrodes are placed over the motor point regions of selected muscles of the lower extremities.

After placement of markers and recording electrodes, the subjects will be instructed to walk down the gait lab runway over the force platform. Simultaneous kinematic, EMG and force plate data is collected. Between 3 and 10 strides of data are collected depending on the degree of variability in the gait pattern. When assistive devices ( canes etc.) or orthotic devices are used, the subject may be asked to ambulate with and without the gait aid.

Since the patients recruited for this study will have abnormalities in their gait, the most significant risk is falling. Therefore, subjects will be screened to ensure that they can ambulate independently over level ground. During testing, standby assistance will be present to help subjects in cases of balance loss. The risks for normal subjects are negligible.

ELIGIBILITY:
Inclusion Criteria:

* Since it is desirable to include the spectrum of gait disorders that are typically encountered in clinical practice, inclusion/exclusion criterion for patients are limited.

Exclusion Criteria:

* Patients must be able to walk independently with or without assistive devices.
* Normal subjects must have no history of neuromuscular or musculoskeletal disorders that interfere with ambulation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults aged 18-75
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 1998-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Gait Parameters | Not a clinical trial. Study closed to enrollment.

SECONDARY OUTCOMES:
Balance | Not a clinical trial. Study closed to enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Walsh, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- South Texas Veterans Healthcare System, San Antonio, Texas, United States